CLINICAL TRIAL: NCT00304460
Title: Studies on the Mechanism of Action of High-Dose IL-2 in Metastatic Melanoma and Renal Cell Cancer
Brief Title: Mechanism of Action of High-Dose IL-2 (Aldesleukin) in Metastatic Melanoma and Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060115; 06-C-0115; NCT00331617 (obsolete NCT alias)
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-02-27

CONDITIONS: Metastatic Melanoma; Renal Cell Cancer
Keywords: Serum Protein Levels; Lymphocyte Phenotypes; Predictive Analysis; Serum Cytokines; Kidney Cancer; Renal Cell Cancer; Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Kidney Neoplasms | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
Background:

-Although IL-2 can shrink tumors in about 20 percent of patients with metastatic kidney cancer and in 15 percent of patients with metastatic melanoma, it is not fully known how the drug works.

Objectives:

-To better understand how IL-2 causes tumors to shrink.

Eligibility:

-Patients 18 years of age or older with metastatic kidney cancer or metastatic melanoma

Design:

* 135 patients with melanoma and 110 patients with kidney cancer may be enrolled.
* Patients are hospitalized for about 7 days for each treatment. They receive IL-2 intravenously (through a vein) over 15 minutes every 8 hours for up to 4 days or 12 doses. This constitutes one treatment cycle.
* Research blood samples are collected daily during the first treatment cycle and for one or two days following the last dose.
* Patients may be asked to undergo leukapheresis, a procedure for collecting large quantities of white blood cells. This involves collecting blood through a needle in an arm vein. The blood is directed through a cell separator where the white cells are extracted. The rest of the blood (red cells, platelets, and plasma) is returned to the patient through the same needle or through a needle in the other arm.
* About 7-10 days after discharge from the hospital, patients return for a second treatment cycle but without research blood sampling.
* 2 months after therapy, patients are evaluated with scans, and x-rays, and blood tests to evaluate the tumor and the effects of the treatment on immune cells.
* Patients whose tumors shrink or remain stable may continue treatment (without repeating the full set of research blood samples) as long as they benefit from the treatment and do not develop unacceptable side effects. Patients who continue treatment are evaluated every 2 months for 3 to 4 times and then every 3 to 6 months.

DETAILED DESCRIPTION:
Background:

* Although interleukin-2 (IL-2) was approved as standard therapy by the US Food and Drug Administration for metastasis melanoma and renal cell carcinoma, the mechanism of action in these patient populations is still not completely understood.
* Methods for studying regulatory T-cells and measuring recently discovered cytokines were not available during earlier studies of IL-2 administration.

Objectives:

- Explore peripheral blood samples of patients with metastatic renal cell cancer or melanoma receiving high-dose IL-2 to identify serum protein levels and lymphocyte phenotypes that may be associated with or predictive of tumor regression.

Eligibility:

* Patients with metastatic renal cell cancer or melanoma who are greater than or equal to 18 years of age, with an ECOG of 0 or 1 who have an expected survival greater than three months.
* Patients with systemic infections, coagulation disorders, or major medical illnesses of the cardiovascular, respiratory or immune system will be excluded, including patients with ejection fractions less than 45% or FEV1 or VC less than or equal to 60% predicted.
* Patients must not have had prior therapy within 28 days, previous IL-2 therapy, be pregnant, have untreated or clinically significant tumor involvement of the CNS or major nerve compression, or have greater than 25% estimated hepatic replacement.

Design:

* Aldesleukin 720,000 IU/kg intravenous bolus over 15 minutes every eight hours for up to 12 doses will be administered as a cycle of treatment.
* Seven to 10 days after discharge, a second cycle of treatment will be administered.
* 20 mLs of blood for serum and 20 mLs of blood for peripheral blood cells will be collected daily during the first cycle of aldesleukin administration and the day following the last dose. 20 mLs of blood for serum and 50 mLs of blood for cell separation will be obtained on days 2 through 4 following completion of IL-2 administration. On one of these days, an additional 50 mLs of blood for cell separation or a 2 hour apheresis may be substituted.
* Approximately two months from the beginning of therapy, a response assessment will be performed.
* Patients with stable or regressing disease will receive a second complete treatment course. Subsequent courses may be administered if there is evidence of on-going tumor regression without long-term or irreversible toxicity.
* In the first 5 patients of each diagnosis (metastatic renal cell cancer and melanoma) the following cytokine levels will be assayed: VEGF, CD40L, FASL, TRAIL, GRO-alpha, IP10, GM-CSF, IFN-gamma, IFN-alpha, IL-1, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-15, TNF-alpha, TNF-beta; and the following phenotypic markers will be studied: CD3, CD4, CD8, CD16, CD25, CD27, CD28, CD56, CD80, CD95, CD107a, CD152, FoxP3, annexin V.
* After the first 10 patients have been analyzed, the scope of the tests will be narrowed to those which show a response to IL-2.
* Initially, a total of 127 evaluable patients with melanoma will be enrolled, with a presumed 15% response rate. With the approval of amendment F, a new accrual ceiling of 200 patients with metastatic melanoma will be established to complete the proposed analysis.
* A total of 100 evaluable patients with renal cell carcinoma will be enrolled with a presumed 20% response rate.
* Allowing for a small number of inevaluable patients, a total of 200 patients with melanoma and 110 patients with renal cell carcinoma may be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any patient with metastatic, measurable, histologically-proven RCC or melanoma who is a candidate for high-dose IL-2 therapy.
* Expected survival greater than three months.
* Age greater than or equal to18 years old.
* ECOG less than 2.
* Serum creatinine less than or equal to 1.4 mg/dl or creatinine clearance greater than or equal to 90 mL/min, and total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
* Platelet count greater than 100,000/mm(3).
* Absolute neutrophil count greater than 1000/mm(3).
* Serum ALT/AST less than three times the upper limit of normal.
* Must be willing to sign a durable power of attorney.
* Must be willing to practice effective contraception (regardless of gender).
* Must be willing to sign the informed consent document.

EXCLUSION CRITERIA:

* Significant second malignancy within 3 years of protocol entry or likely to require intervention in the year following protocol entry.
* Significant psychiatric disease which in the opinion of the Principal Investigator would prevent adequate informed consent or render immunotherapy unsafe or contraindicated.
* Requirement for systemic or inhaled steroid administration (topical therapy is acceptable).
* Prior therapy within 28 days (except focal radiation for bone lesion).
* Systemic infections, coagulation disorders or evidence of active bleeding, or other major medical illnesses of the cardiovascular, respiratory or immune system.
* ECOG performance status greater than 2.
* Pregnancy.
* Previous IL-2 therapy.
* Positive HIV antibody titer, Seropositive for hepatitis B or C antigen.
* FEV1 or VC less than or equal to 65% of predicted (pulmonary function screening to be done in patients with significant smoking history [greater than 20pk/years] or suspicion of pulmonary disease by history or examination).
* Abnormal stress cardiac exam (to be done in all patients greater than or equal to 60 years old and others as indicated clinically) or active cardiac ischemia or significantly abnormal EKG.
* Greater than 25% estimated hepatic replacement by tumor or SGOT or SGPT greater than 3x normal.
* Untreated or clinically significant (i.e. because of size or presence of edema) tumor involvement of the CNS or major nerve compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2006-03-13; Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

PRIMARY OUTCOMES:
Clinical outcome as measured by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: James C Yang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rigel DS, Carucci JA. Malignant melanoma: prevention, early detection, and treatment in the 21st century. CA Cancer J Clin. 2000 Jul-Aug;50(4):215-36; quiz 237-40. doi: 10.3322/canjclin.50.4.215. PMID 10986965
- [Background] Lin JX, Leonard WJ. Signaling from the IL-2 receptor to the nucleus. Cytokine Growth Factor Rev. 1997 Dec;8(4):313-32. doi: 10.1016/s1359-6101(97)00021-x. PMID 9620644
- [Background] Koizumi S, Seki H, Tachinami T, Taniguchi M, Matsuda A, Taga K, Nakarai T, Kato E, Taniguchi N, Nakamura H. Malignant clonal expansion of large granular lymphocytes with a Leu-11+, Leu-7- surface phenotype: in vitro responsiveness of malignant cells to recombinant human interleukin 2. Blood. 1986 Nov;68(5):1065-73. PMID 2945603